CLINICAL TRIAL: NCT00001106
Title: A Phase I Trial To Evaluate Zidovudine (ZDV) in HIV-1 Infected Pregnant Women and Their Offspring
Brief Title: A Study of Zidovudine in HIV-Infected Pregnant Women and Their Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 082; 11057 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Pregnancy
Keywords: Pregnancy; Pregnancy Complications, Infectious; Prenatal Exposure Delayed Effects; Drug Evaluation; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious; Prenatal Exposure Delayed Effects; Acquired Immunodeficiency Syndrome | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
AMENDED: To evaluate the pharmacokinetics of intravenously administered AZT to HIV-1 infected pregnant women in labor; to evaluate the pharmacokinetics and urinary excretion of AZT and its metabolites in newborns of HIV-1 infected mothers who receive IV AZT only during labor; to evaluate the safety of IV AZT administered by continuous infusion to HIV-1 infected laboring women and their infants. Original design: To determine the distribution and elimination of zidovudine (AZT) in the body as well as its safety in the treatment of pregnant women and their unborn children. The information derived from this study is required in order to design a future study that will assess the efficacy of AZT in reducing the transmission rate of HIV-1 from seropositive women to their fetus by treating them during the third trimester of pregnancy.

An estimated 30 percent to 40 percent infected pregnant women risk transmission of HIV-1 to their infants, whether they be symptomatic or asymptomatic. Zidovudine (AZT) has previously demonstrated its effectiveness as a potent inhibitor of HIV replication in vitro and in adult patients; benefits of treatment include decreased mortality rate, decreased incidence of opportunistic infections, and increased number of CD4 cells. Phase I AZT studies in children, however, have resulted in uncontrolled information regarding clinical efficacy. The present study, therefore, will investigate the safety and pharmacokinetics of intravenous (IV) and oral AZT administration to HIV-1 infected pregnant women in the 3rd trimester, as well as the safety and efficacy of such treatment in their newborns.

It is hoped that the results will be instrumental in designing future studies to assess the efficacy of AZT in reducing the transmission risk of HIV-1.

DETAILED DESCRIPTION:
An estimated 30 percent to 40 percent infected pregnant women risk transmission of HIV-1 to their infants, whether they be symptomatic or asymptomatic. Zidovudine (AZT) has previously demonstrated its effectiveness as a potent inhibitor of HIV replication in vitro and in adult patients; benefits of treatment include decreased mortality rate, decreased incidence of opportunistic infections, and increased number of CD4 cells. Phase I AZT studies in children, however, have resulted in uncontrolled information regarding clinical efficacy. The present study, therefore, will investigate the safety and pharmacokinetics of intravenous (IV) and oral AZT administration to HIV-1 infected pregnant women in the 3rd trimester, as well as the safety and efficacy of such treatment in their newborns.

It is hoped that the results will be instrumental in designing future studies to assess the efficacy of AZT in reducing the transmission risk of HIV-1.

AMENDED: For the pharmacokinetic and safety study of AZT during labor and in the newborn infants, women who were screened and have consented are included in this part of the study. 6 mother-infant pairs without a history of intravenous drug abuse and 4 pairs with such a history are evaluated. The mother receives an infusion of AZT over 1 hour followed by continuous infusion of AZT for at least 4 hours until delivery. Pharmacokinetic data is collected on all patients including those who deliver before receiving 4 hours of AZT infusion.

AMENDED: The trial will proceed as described above except that the first 2 methadone patients enrolled will receive half the AZT dose given to the non-methadone patients. Results will be evaluated before dosing of additional methadone-use patients is done. Original design: Following evaluation, patients receive one intravenous dose of AZT over a 1-hour period. One day later, patients begin taking AZT capsules 5 times a day by mouth for the remaining weeks prior to labor.

During labor, patients continue to receive AZT intravenously every 4 hours until they deliver their babies. Blood and urine tests are made to measure the amounts of AZT in the mother's and, after delivery, the baby's body fluids. AZT is stopped after the baby has been delivered. The initial enrollment is six women with no history of intravenous drug abuse plus another four women with a history of intravenous drug use, who have been receiving methadone maintenance therapy. These women are not required to have a negative urine toxicology screen for illicit drugs to enter the study.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* In one group of four or more patients, methadone maintenance treatment.
* Acetaminophen for periods less than 72 hours.
* Supportive therapy including blood and blood products, vaginal creams, antiemetics, antidiarrheals, and cough medicines as deemed necessary by the responsible investigator.
* Iron, multivitamins, and short course of treatment for correctable medical problems, such as urinary tract infection.

Concurrent Treatment:

Allowed:

* Blood and blood products as supportive therapy.

Patients must have HIV-1 infection and be in the third trimester of pregnancy. Additional patients will also be receiving methadone maintenance therapy for intravenous drug use.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Systemic medications during this pregnancy.
* Acetaminophen for periods more than 72 hours.

Patients will be excluded from the study for the following reasons:

* Complications of pregnancy.
* History of poor medical compliance related to factors other than accessibility of care.
* Insistence on breast-feeding during the first 24 hours of the birth of the child.
* Evidence of preexisting fetal anomalies at = or > 20 weeks gestation as noted by an abnormal level 2 sonogram prior to study entry.
* Evidence of fetal intolerance of the intrauterine environment including intrauterine growth retardation, oligohydramnios, polyhydramnios, biophysical profile equal to or less than 6 for fetus with a gestational age > 32 weeks, congenital malformation, fetal hydrous or ascites.
* Previous systemic infection including influenza during this pregnancy.
* Malabsorption syndrome and/or history of frequent diarrhea that might interfere with absorption of oral zidovudine (AZT).

Prior Medication:

Excluded:

* Antivirals and other systemic medications during this pregnancy.

Patients may not have any of the following diseases or symptoms:

* Obstetrical complications:
* Poor obstetrical history including but not limited to recurrent spontaneous abortions, previous preterm or low-birth-weight infant, congenital anomalies (past or present pregnancy), premature rupture of membranes, multiple gestation, intrauterine fetal death (this pregnancy), and placenta previa or abruptio (this pregnancy).
* Medical complications:
* Conditions including but not limited to insulin-dependent diabetes mellitus (IDDM), hypertensive disorders which include preeclampsia, eclampsia, chronic hypertension, cardiovascular disease including rheumatic or congenital heart disease, collagen vascular disease, endocarditis, and renal disease.
* Hematologic complications.
* Neurologic complications.
* Pulmonary complications.

History of illicit drug use during this pregnancy.

* Note: This exclusion applies only to the first six or more women to enter this study who do not have a history of intravenous drug use.

Four or more patients:

* Intravenous drug use, if enrolled in a methadone maintenance program.

Ages: 1 Day to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40
Dates: Study Completion 1994-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: O'Sullivan MJ, Study Chair; Parks W, Study Chair
Locations (9):
- United States (9):
  - Kaiser - Edgemont Street / UCLA Med Ctr, Los Angeles, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - Univ of Miami (Pediatric), Miami, Florida
  - Boston City Hosp / Pediatrics, Boston, Massachusetts
  - UMDNJ - New Jersy Med School, Newark, New Jersey
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Children's Hosp of Seattle, Seattle, Washington
  - Univ of Washington, Seattle, Washington